CLINICAL TRIAL: NCT06572709
Title: Ultrasonographic Evaluation of Parasternal Intercostal Muscles and Their Correlation With Respiratory Function Test in Stroke Patients
Brief Title: Ultrasonographic Evaluation of Parasternal Intercostal Muscles in Stroke Patients
Acronym: UEPIMSP
Status: Recruiting | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FSMYED
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Stroke; Respiratory Muscle
Keywords: stroke; intercostal muscle; pulmonary function test; respiratory muscle; ultrasound
MeSH Terms: conditions — Stroke | interventions — Ultrasonography; Spirometry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke patients: Ultrasonographic measurements were performed of the bilateral parasternal intercostal muscle thickness. Spirometry evaluation was performed by another investigator.
  Interventions: Diagnostic Test: Parasternal intercostal muscle thickness with ultrasonography
- Healthy individuals: Ultrasonographic measurements were performed of the dominant side parasternal intercostal muscle thickness. Spirometry evaluation was performed by another investigator.
  Interventions: Diagnostic Test: Parasternal intercostal muscle thickness with ultrasonography

INTERVENTIONS:
Diagnostic Test: Parasternal intercostal muscle thickness with ultrasonography — Ultrasonographic measurements were performed of the bilateral parasternal intercostal muscle thickness in the supine position in the stroke patient group. Ultrasonographic measurements were performed of dominant side parasternal intercostal muscle thickness in the supine position in healthy individuals group. Spirometry evaluation was performed in both groups.
  Other Names: Spirometry

SUMMARY:
Ultrasonographic evaluation of parasternal intercostal muscles and to determine whether there is a correlation with PFT parameters in stroke patients

DETAILED DESCRIPTION:
The clinical study, planned as a cross-sectional prospective, will be conducted on 30 stroke patients followed in the same stroke clinic and a total of 30 healthy volunteers of similar age and gender to the stroke patients. Patients with ischemic or hemorrhagic stroke with stroke duration >6 months and mini-mental test score >24 will be included in the study; Stroke patients with acute or chronic lung disease, a history of thoracic surgery, another neuromuscular disease, aphasia type in which comprehension is impaired, and facial paralysis will not be included in the study. Written informed consent will be obtained from those who meet the study criteria and agree to participate in the study.

Demographic data of patients and healthy volunteers (gender, age, height, weight, body mass index, dominant extremity, stroke etiology, duration, side), respiratory function test (PFT) parameters measurement results, bilateral parasternal intercostal muscle thickness in stroke patients and the dominant side parasternal intercostal muscle thicknesses in healthy volunteers will be measured with Ultrasound (US), thickening rates will be calculated and recorded.

All participants will be evaluated in B-mode using the MyLab60 brand US device with 7-12 MHz linear probe. Measurements will be taken at the end of tidal expiration and maximal inspiration while the participants are in the supine position. To evaluate intercostal muscle thickness, measurements will be made between the 2nd and 3rd ribs, 3 cm lateral to the sternum, in accordance with the literature. The probe will be placed vertically at this point in the sagittal plane, a vertical caliper will be drawn between the hyperechoic fascia lines on the pleura and this distance will be recorded in millimeters. All measurements will be repeated 3 times, the average value will be recorded and thickening rates will be calculated. The formula [(end-inspiratory thickness - end-expiratory thickness) / end-expiratory thickness] will be used to calculate the thickening ratio. US evaluation of each participant will be performed by an experienced physician with more than 5 years of experience in this field.

Respiratory functions of the individuals included in the study will be measured with a CHEST HI-105 10510759 model spirometer, according to the American Thoracic Society and European Respiratory Society criteria. Forced vital capacity [FVC], forced expiratory volume in 1 second [FEV1], FEV1/FVC, maximal expiratory flow rate [PEF] values and their percentage predictive values will be recorded. MicroRPM Respiratory Meter device (MicroDirect, USA) will be used for respiratory muscle strength measurements (maximum inspiratory pressure [MIP] maximum expiratory pressure [MEP]). PFT of all participants will be performed by a different researcher who is blind to the US measurement results.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or Hemorrhagic stroke patients, Stroke duration >6 months, Mini-mental test score >24

Exclusion Criteria:

* Individuals with acute or chronic lung disease, Patients with a history of thoracic or abdominal surgery, Patients with other neuromuscular diseases, Aphasia type with impaired understanding, Facial paralysis

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stroke patients and healthy volunteers (have close demographic data with stroke patients)
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2024-08-28 (Estimated); Study Completion 2024-09-04 (Estimated)

PRIMARY OUTCOMES:
Parasternal intercostal muscle thickness and thickening ratio | 15 minute
  Parasternal intercostal muscle ultrasonographic millimetric measurement

SECONDARY OUTCOMES:
Correlation between parasternal intercostal muscle thicknesses and spirometry parameters | 15 minute
  Vital capacity[VC], forced vital capacity [FVC], forced expiratory volume 1 second [FEV1] , FEV1/FVC, maximal expiratory flow rate [PEF], maximum inspiratory pressure [MIP] maximum expiratory pressure [MEP] in patients' PFT ]

CONTACTS AND LOCATIONS:
Overall Officials: Yunus Emre Dogan, MD, Principal Investigator — Istanbul Fatih Sultan Mehmet Training and Research Hospital; Kadriye Ones, Prof, Study Chair — Istanbul Physical Medicine Rehabilitation Training and Research Hospita; Cigdem Cinar, Assoc Prof, Study Chair — Istanbul Biruni University; Burak Kutuk, MD, Study Chair — Hatay Defne State Hospital; Muhsin Doran, MD, Study Chair — Isttanbul Liv Hospital
Locations (1):
- Istanbul Physıcal Therapy And Rehabılıtatıon Traınıng And Research Hospıtal, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wallbridge P, Parry SM, Das S, Law C, Hammerschlag G, Irving L, Hew M, Steinfort D. Parasternal intercostal muscle ultrasound in chronic obstructive pulmonary disease correlates with spirometric severity. Sci Rep. 2018 Oct 15;8(1):15274. doi: 10.1038/s41598-018-33666-7. PMID 30323179
- [Background] Yoshida R, Tomita K, Kawamura K, Nozaki T, Setaka Y, Monma M, Ohse H. Measurement of intercostal muscle thickness with ultrasound imaging during maximal breathing. J Phys Ther Sci. 2019 Apr;31(4):340-343. doi: 10.1589/jpts.31.340. Epub 2019 Apr 1. PMID 31037006
- [Background] Formenti P, Umbrello M, Dres M, Chiumello D. Ultrasonographic assessment of parasternal intercostal muscles during mechanical ventilation. Ann Intensive Care. 2020 Sep 7;10(1):120. doi: 10.1186/s13613-020-00735-y. PMID 32894372
- [Background] Yoshida R, Tomita K, Kawamura K, Setaka Y, Ishii N, Monma M, Mutsuzaki H, Mizukami M, Ohse H, Imura S. Investigation of inspiratory intercostal muscle activity in patients with spinal cord injury: a pilot study using electromyography, ultrasonography, and respiratory inductance plethysmography. J Phys Ther Sci. 2021 Feb;33(2):153-157. doi: 10.1589/jpts.33.153. Epub 2021 Feb 13. PMID 33642691